CLINICAL TRIAL: NCT05355987
Title: Impact of Point in Time of Introducing Paramedical Consultations in Oncological Supportive Care in Outpatients With Multiple Myeloma
Brief Title: Impact of Paramedical Consultations in Oncological Supportive Care in Outpatients With Multiple Myeloma
Acronym: SOSAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHB21.01
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: supportive care; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early oncological supportive care (Experimental): Evaluation of needs in oncological supportive care by a nursing coordinator from diagnosis and recommendation to plan appointments with different specialists in supportive care regarding to patient's needs
  Interventions: Other: Early oncological supportive care
- Delayed oncological supportive care (Other): Evaluation of needs in oncological supportive care by a nursing coordinator at 6 months after diagnosis and recommendation to plan appointments with different specialists in supportive care regarding to patient's needs
  Interventions: Other: Delayed oncological supportive care

INTERVENTIONS:
Other: Early oncological supportive care — Several appointments (at diagnosis, 3 months, 6 months and 9 months) with nursing coordinator to define the needs in oncological supportive care. Different appointments will be planned according to patient's needs, with several possibilities: oncological supportive care nurse, social worker, psychologist, physiotherapist, adapted physical activity, medication reconciliation, oncologic geriatric medicine, dietician, nutritionist, smoking cessation advisor, sexologist, sophrologist, pain management nursing and palliative care, socio-aesthetician and religious cult coordinator.
  Arms: Early oncological supportive care
Other: Delayed oncological supportive care — Two appointments (6 months and 9 months) with nursing coordinator to define the needs in oncological supportive care. Different appointments will be planned according to patient's needs, with several possibilities: oncological supportive care nurse, social worker, psychologist, physiotherapist, adapted physical activity, medication reconciliation, oncologic geriatric medicine, dietician, nutritionist, smoking cessation advisor, sexologist, sophrologist, pain management nursing and palliative care, socio-aesthetician and religious cult coordinator.
  Arms: Delayed oncological supportive care

SUMMARY:
Multiple myeloma is the second most frequent hematologic malignancy, which incidence augmented between 1995 and 2018, with an annual mean variation of +0.6% to 1.1%. Although treatment improved in the last years, the patients' prognostic is associated with cytogenetic abnormalities.

Oncological supportive care provides patients with a global perspective, in addition to specific medical treatment adapted to pathology and patient profile. It contributes to the improvement of quality of life of patients, throughout their care pathway regarding physical, psychological and social aspects, according to their specific needs as well as their caregivers'.

The aim of this study is to evaluate the quality of life at 6 months after multiple myeloma diagnosis in outpatients receiving paramedical consultations in oncological supportive care from the diagnosis versus outpatients receiving paramedical consultations in oncological supportive care after 6 months after diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age superior to 18 years old
* Patient recently diagnosed with multiple myeloma not eligible to autologous blood stem-cell transplantation, before starting therapy in day hospital
* Patient coming regularly to Centre Henri Becquerel for treatment and follow up for multiple myeloma
* Informed consent form signed

Exclusion Criteria:

* Inclusion Criteria:
* Age superior to 18 years old
* Patient recently diagnosed with multiple myeloma not eligible to autologous blood stem-cell transplantation, before starting therapy in day hospital
* Patient coming regularly to Centre Henri Becquerel for treatment and follow up for multiple myeloma
* Informed consent form signed

Exclusion Criteria:

* Patient with urgent need of treatment after multiple myeloma diagnosis with urgent and absolute need of oncological supportive care immediately after diagnosis
* Patient deprived of liberty, under judicial supervision, under guardianship or trusteeship
* History of psychological or sensorial disorder or anomaly that can prevent the patient from understanding the conditions for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Comparison of quality of life evolution in outpatients with multiple myeloma between the two groups | 6 months
  Comparison of the score obtained with Functional Assessment of Cancer Therapy- Multiple Myeloma questionnary

SECONDARY OUTCOMES:
Qualitative evaluation of quality of life | 6 months
  Semi-structured individual interviews
Comparison of quality of life in outpatients with multiple myeloma between the two groups | 3 months
  Comparison of the score obtained with Functional Assessment of Cancer Therapy- Multiple Myeloma questionnary
Comparison of quality of life in outpatients with multiple myeloma between the two groups | 9 months
  Comparison of the score obtained with Functional Assessment of Cancer Therapy- Multiple Myeloma questionnary
Comparison of autonomy evolution in outpatients with multiple myeloma between the two groups | 6 months
  Comparison of the score of Instrument Activities of daily Living questionnary

CONTACTS AND LOCATIONS:
Overall Officials: Amel Benchemam, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No